CLINICAL TRIAL: NCT04633161
Title: The Role of Quadriceps and Hamstring Muscles in Knee Stability During Single Leg Hop Landing in Patients With Anterior Cruciate Ligament Reconstruction
Brief Title: The Role of Muscle in Knee Stability
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Xin He, PhD candidate, Chinese University of Hong Kong
Other Study IDs: 2019.100
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: muscle strength; muscle elasticity; muscle coordination; knee stability
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to compare the difference in muscle strength, muscle elasticity and muscle coordination of quadriceps and hamstring muscle and their association with knee biomechanics during single leg hop landing in patients with anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
In Hong Kong, over 3000 cases of Anterior Cruciate Ligament Reconstruction (ACLR) are operated annually to restore knee stability. Despite recovery of knee passive laxity and muscle strength, dynamic knee stability is often not restored. In additional to muscle strength, muscle elasticity and muscle coordination may also play an important role in knee stability. However, there is no evidence regarding the changes in muscle elasticity after ACLR and its contribution to dynamic knee stability. This study is a cross-sectional study designed to compare the the difference in muscle strength, muscle elasticity and muscle coordination of quadriceps and hamstring muscle in 30 ACLR patients and investigate its relationship with knee biomechanics during single leg hop landing. Patient selection was base on medical records and subjective knee functional scores. Patient enrollment and informed consent was conducted first. Muscle strength was measured by isokinetic muscle testing(Biodex) at two speeds. Muscle elasticity was assessed by ultrasound shear wave elastography. Muscle coordination evaluated by electromyography(EMG) and knee biomechanics including kinematics and kinetics was measured by 3D motion analysis system(VICON) and all the assessments were done in CUHK-ORT Sports Injury Research Laboratory in the Prince of Wales Hospital, Hong Kong. All data was collected and analyzed by qualified personnel.

ELIGIBILITY:
Inclusion Criteria:

* (1) Male aged 18-35 (2) With pre-injury activity level of more than 6 in Tegner score (3) Within their post-operative 6-18 months (4) Without injury history for the contralateral limb

Exclusion Criteria:

* (1) With concomitant fracture, meniscus injury or chondral lesion (2) With preoperative radiographic signs of arthritis (3) With revision ACL surgery (4) With injury history of the spine or hamstring strain during the past 6 months.

Ages: 18 Years to 35 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes — based on self-report of gender identity
Study Population: Young and active ACL patients within their post-ACLR 6-18 months
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
knee biomechanics during single leg hop landing | post-operatively 6-18 months
  knee kinematics(peak knee flexion, knee valgus, knee internal rotation, knee flexion excursion, valgus excursion and internal excursion) and kinetics(vertical ground reaction force, knee extension moment, knee valgus moment) were collected by 3D motion analysis system(VICON) during the landing phase of single leg hop test
muscle strength | post-operatively 6-18 months
  muscle peak torque of knee extension and knee flexion at 60°/s and 180°/s tested with isokinetic mode by Biodex
muscle elasticity | post-operatively 6-18 months
  muscle shear elastic modulus of vastus medialis, rectus femoris, vastus lateralis, semimembranosus,semitendinosus and biceps femoris was measured by ultrasound shear wave elastography
muscle coordination | post-operatively 6-18 months
  muscle activity level and onset time of vastus medialis, vastus lateralis, semimembranosus,and biceps femoris was assessed by electromyography(EMG) during the landing phase of single leg hop test

SECONDARY OUTCOMES:
knee laxity | post-operatively 6-18 months
  anterior displacement of the tibia was measured using the KT-1000 arthrometerat 134 N with knee flexed at around 20°
subjective knee function | post-operatively 6-18 months
  International Knee Documentation Committee (IKDC) scoring system, which is consisted of 10 questions about symptoms and activity ranging from 0 to 100
Psychological readiness for return-to-play | post-operatively 6-18 months
  Anterior Cruciate Ligament-Return to Sport after Injury(ACL-RSI)-on a scale from 0 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- The chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided